CLINICAL TRIAL: NCT02582372
Title: Subarachnoidal Anesthesia: Dexmedetomidine vs Fentanyl Plus Hyperbaric Bupivacaine for Lower Abdomen Surgery
Acronym: Dex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Central Dr. Luis Ortega (Other)
Responsible Party: Principal Investigator, Beatriz Arismendi Gómez, Clinical Professor Beatriz Arismendi Gomez, Hospital Central Dr. Luis Ortega
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCLuisOrtega
Record Dates: First submitted 2015-10-07; First posted 2015-10-21 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Dexmedetomidine in Subarachnoidal Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine (Experimental): 25 patients recieve subarachnoidal anesthesia with 12,5 mgrs of bupivacaine 0,5% plus 10 micrograms of dexmedetomidine, with needle 25 gauge
  Interventions: Drug: Dexmedetomidine and bupivacaine
- fentanyl (Active Comparator): 25 patients recieve subarachnoidal anesthesia with 12,5 mgrs of bupivacaine 0,5% plus 25 micrograms of fentanyl, with needle 25 gauge
  Interventions: Drug: Fentanyl and bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine and bupivacaine — 10 micrograms of dexmedetomidine plus 12,5 mgrs of bupivacaine subarachnoideal
  Arms: dexmedetomidine
Drug: Fentanyl and bupivacaine — 25 micrograms of fentanyl plus 12,5 mgrs of bupivacaine subaracnoideal
  Arms: fentanyl

SUMMARY:
Dexmedetomidine, highly selective agonist for alpha-2 receptors, enhances the sensory and motor block with prolonged postoperative analgesia without hemodynamic compromise.

OBJECTIVE: To evaluate effects of dexmedetomidine vs fentanyl with hyperbaric bupivacaine spinal anesthesia for lower abdominal surgeries.

METHODS: double-blind, randomized, American Society Anesthesiologist classification (ASA) : I - II, 18-65 years. F group (23 patients) received 25 mcg fentanyl, Group D (27 patients), 10 mcg dexmedetomidine with 12.5 mg hyperbaric bupivacaine . 0,02mgrs morphine / kg intravenously if EVA≥4was administered in postoperative period. Hemodynamic variables and O2 saturation intraoperatively was recorded, EVA every 4 hours, side effects, sensory block, motor, sedation and peripheral neurological manifestations of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* lower abdominal surgery

Exclusion Criteria:

* Consumption antagonists adrenergic or channel blockers Ca ++
* Patients with arrhythmias or heart block
* Allergic to any drugs under study
* Obese
* Physical or mental incapacity to understand and use the pain scale
* Contraindication for anesthesia conductive
* Realization difficulty or complication during anesthesia and / or surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes of baseline blood pressure | during anesthesia and 1 hour of postoperatory
Changes of baseline cardiac rate | during anesthesia and 1 hour of postoperatory
Changes of baseline oxygen saturation | during anesthesia and 1 hour of postoperatory
Postoperatory pain visual analogue scale | during first 24 hours of postoperatory
Changes of motor block using Bromage scale | during anesthesia and 1 hour of postoperatory

SECONDARY OUTCOMES:
Numbers of patients with hypotension using non invasive blood presure monitor | during anesthesia and first 24 hours of postoperatory
  we report hypotension below 20% of basal values
Numbers of patients with excessive sedation using Ramsay scale | during anesthesia and first 24 hours of postoperatory
Numbers of patients with nauseas | during anesthesia and first 24 hours of postoperatory

OTHER OUTCOMES:
Numbers of patients with signs of peripheral neurological toxicity using questionnaire | during first seven days of postoperatory time
  phone contact